CLINICAL TRIAL: NCT04364802
Title: Povidone-Iodine Intranasal for Prophylaxis in Front-line Health-care Personnel and Inpatients During the Sars-CoV-2 Pandemic
Brief Title: COVID-19: Povidone-Iodine Intranasal Prophylaxis in Front-line Healthcare Personnel and Inpatients
Acronym: PIIPPI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nikita Gupta (Other)
Responsible Party: Sponsor-Investigator, Nikita Gupta, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 58748
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: COVID-19; SARS-CoV 2
Keywords: COVID-19; SARS-CoV 2; Health Care Workers; COVID-19 Prophylaxis
MeSH Terms: conditions — COVID-19 | interventions — Mouthwashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Healthcare Workers - Control (No Intervention): Front-line healthcare workers (FLCHW) who are negative for COVID will receive standard PPE and a pre- and post-study test for COVID-19.
- Healthcare Workers - PVP-I (Experimental): Front-line healthcare workers (FLCHW) who are negative for COVID-19 will receive standard PPE and a pre- and post-study test for COVID-19. Additionally, they will receive PVP-I spray and gargle.
  Interventions: Drug: Povidone-Iodine Nasal Spray and Gargle
- Inpatients - Control (No Intervention): Inpatients who have a 7+ day hospitalization or who are set to undergo a significant surgical procedure will receive standard care and a pre- and post-study COVID-19 test.
- Inpatients - PVP-I (Experimental): Inpatients who have a 7+ day hospitalization or who are set to undergo a significant surgical procedure will receive standard care and a pre- and post-study COVID-19 test. Additionally, they will receive PVP-I gargle and nasal sprays that will be applied shortly after admission or perioperatively.
  Interventions: Drug: Povidone-Iodine Nasal Spray and Gargle
- Community - Control (No Intervention): Community participants who are negative for COVID-19 will receive a pre- and post-study COVID-19 test.
- Community - PVP-I (Experimental): Community participants who are negative for COVID-19 will receive a pre- and post-study COVID-19 test. Additionally, they will receive PVP-I gargle and nasal sprays.
  Interventions: Drug: Povidone-Iodine Nasal Spray and Gargle

INTERVENTIONS:
Drug: Povidone-Iodine Nasal Spray and Gargle — Healthcare workers will receive standard PPE and a pre- and post-study nasal swab COVID19 test. Additionally, they will receive povidone-iodine nasal spray and gargle (10% diluted 1:30) to use at the beginning of their shift, in the middle, and at the end of their shift.
  Arms: Healthcare Workers - PVP-I
Drug: Povidone-Iodine Nasal Spray and Gargle — Patients will receive standard of care treatment and a pre- and post-study nasal spray COVID19 test. Additionally, they will receive povidone-iodine nasal spray and gargle shortly after admission or preoperatively.
  Arms: Inpatients - PVP-I
Drug: Povidone-Iodine Nasal Spray and Gargle — Community members will receive a pre- and post-study nasal swab COVID19 test. Additionally, they will receive povidone-iodine nasal spray and gargle (10% diluted 1:30) to use at home.
  Arms: Community - PVP-I

SUMMARY:
Povidone-iodine (PVP-I) is a broad-spectrum antiseptic with activity against bacteria, fungi, and viruses. It has been previously used in both intranasal preparations against Methicillin Resistant Staphylococcus Aureus (MRSA) as well as oral preparations in in-vitro studies of Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV), Middle Eastern Respiratory Syndrome Coronavirus (MERS-CoV), influenza H1N1, and rotavirus with good efficacy. This study will evaluate the efficacy of PVP-I as prophylaxis in Coronavirus Disease 2019 (COVID19)-negative front-line health care workers, hospital patients, and community members.

DETAILED DESCRIPTION:
The COVID-19 pandemic, caused by Severe Acute Respiratory Syndrome Coronavirus - 2 (SARS-CoV-2), has been implicated in over 12 million cases and counting in the United States alone and has killed at least 1300 health care workers and >250,000 citizens. This, added to the national shortage of personal protective equipment (PPE) and the need to reuse PPE, lends to the significantly increased risk to healthcare providers. At the beginning of this trial, there were only 360,000 cases.

The highest concentration of viral particles resides within the nasopharynx. The virus is thought to spread via respiratory droplets with the potential for transmission via inhalation of droplets, contact to the nose and mouth with infected materials, and airborne transmission. Given that frontline workers are involved in high-risk procedures including intubation, bronchoscopy, proning patients (which can lead to droplet production) and in some cases are reusing PPE, finding ways to reduce viral load or viral exposure are paramount.

Povidone-iodine (PVP-I) is a broad-spectrum antiseptic with activity against bacteria, fungi, and viruses. It has been previously used in both intranasal preparations against MRSA as well as oral preparations in in-vitro studies of SARS-CoV-2, MERS-CoV, H1N1, and rotavirus with good efficacy.

Due to the known breadth of its antiviral activity and similarities in molecular structure, it can be extrapolated that PVP-I should have robust activity against SARS-CoV-2. Eggers et al found that at a concentration of 1% there was a reduction of viral activity of 99.99% in in-vitro assays. At 2 minutes, a concentration of 0.23% was enough to reduce viral loads appreciably. New data has demonstrated efficacy in-vitro of PVP-I against SARS-CoV-2 at low concentrations.

PVP-I is widely used as an antiseptic and is well-tolerated and has been shown to have little to no effect on mucociliary clearance, olfaction, or thyroid function if iodine holidays are taken, although care must be utilized in monitoring.

In this study, front line healthcare workers will be asked to complete a pre-participation survey and screened for COVID positivity. They will then be given premade PVP-I gargles and nasal sprays, as well as a calendar card to mark compliance. PVP-I nasal spray and gargle (10% diluted 1:30) will be used prior to the start of a shift, during "lunch break", and at the end of shift. First, the nasal spray will be sprayed in the nose (2 sprays each naris). For adequate coverage, the participant should be able to taste the iodine or see it in the back of the throat. This should be left in place for 30 seconds. Then, the participant will gargle the solution for 30 seconds and not have anything to eat or drink by mouth for 30 minutes. Treatment will continue for 3 weeks, or until the healthcare worker presents with COVID symptoms. Participants will then be tested for COVID positivity and asked to fill out a second questionnaire assessing study tolerability. At completion of the study, they will be asked to turn in their calendar card to assess how many applications they were able to complete.

Given the high rate of asymptomatic carriers, a second arm will also be planned for patients who have a 7+ day hospitalization or who are set to undergo a significant surgical procedure. These patients will be offered participation in the study as well and will be given the same questionnaire and undergo preoperative testing if they consent. For patients in the study group, PVIP gargle and nasal sprays will be applied preoperatively or shortly after admission and enrollment in the study for the non-operative group. The patients will then be retested in 2 weeks or as directed by the presentation of symptoms concerning for infection with SARS-CoV-2.

Community spread has been found to be the most likely implicated in infection and thus the trial is now being expanded to include community members. Thus, a THIRD arm has now been added to include community members. Prescreening questionnaires will be given. As long as the participant has had no prior history of a positive COVID-19 test, they will be considered eligible for participation. After a screening consultation, they will undergo a COVID-19 test (should be completed within 72 hours of screening). If negative, they will be eligible. Participants who are pregnant, breastfeeding, have thyroid disease or cancer, or who have an allergy to iodine/shellfish/or contrast dye can still participate but will automatically be on the control arm. Participants may opt to be on either the PVP-I arm or the control arm. They will be asked to fill out a daily questionnaire regarding their exposures and whether they were wearing a mask or if other people were wearing a mask at that time.

ELIGIBILITY:
Inclusion Criteria:

* healthcare worker OR
* patient with expected hospital stay of 7+ days OR
* patient admitted for major surgery OR
* community member
* COVID19 negative by nasal swab test
* asymptomatic for COVID19
* able to consent

Exclusion Criteria:

* positive for COVID19 by nasal swab
* symptomatic for COVID19
* unable to consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra E Kejner, MD, Principal Investigator — Univesity of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burton MJ, Clarkson JE, Goulao B, Glenny AM, McBain AJ, Schilder AG, Webster KE, Worthington HV. Use of antimicrobial mouthwashes (gargling) and nasal sprays by healthcare workers to protect them when treating patients with suspected or confirmed COVID-19 infection. Cochrane Database Syst Rev. 2020 Sep 16;9(9):CD013626. doi: 10.1002/14651858.CD013626.pub2. PMID 32936949

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthcare Workers - Control | Healthcare Workers - PVP-I | Inpatients - Control | Inpatients - PVP-I | Community - Control | Community - PVP-I
Started | 11 | 38 | 17 | 14 | 2 | 16
Completed | 11 | 38 | 17 | 14 | 2 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthcare Workers - Control | Healthcare Workers - PVP-I | Inpatients - Control | Inpatients - PVP-I | Community - Control | Community - PVP-I | Total
Number analyzed (Participants) | 11 | 38 | 17 | 14 | 2 | 16 | 98
Age, Customized [Mean (Full Range); unit: years]
  Age | 36 [27 to 54] | 41 [23 to 83] | 60 [30 to 79] | 64 [36 to 81] | 61 [52 to 70] | 43 [22 to 72] | 49 [22 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 20 | 6 | 5 | 2 | 9 | 48
  Male | 5 | 18 | 11 | 9 | 0 | 7 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 2 | 4
  Not Hispanic or Latino | 11 | 35 | 14 | 14 | 2 | 13 | 89
  Unknown or Not Reported | 0 | 2 | 2 | 0 | 0 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 5 | 0 | 0 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 0 | 0 | 3
  White | 10 | 30 | 16 | 14 | 2 | 14 | 86
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 38 | 17 | 14 | 2 | 16 | 98

OUTCOME MEASURES:

1. Primary Outcome: Percent of Healthcare Workers Testing Positive for COVID-19.
Description: Percent of healthcare workers that become positive for COVID-19 during the study.
Time Frame: 3 weeks
Population: This outcome measure pertains only to the arms that include healthcare workers.
Measure: Number; unit: percentage of healthcare workers
Arm/Group | Healthcare Workers - Control | Healthcare Workers - PVP-I | Inpatients - Control | Inpatients - PVP-I | Community - Control | Community - PVP-I
Number analyzed (Participants) | 11 | 38 | 0 | 0 | 0 | 0
percentage of healthcare workers | 0 | 0 |  |  |  |

2. Primary Outcome: Percent of Patients Testing Positive for COVID-9.
Description: Percent of patients that become positive for COVID-19 during the study.
Time Frame: 2 weeks
Population: Percentage of patients that become positive for COVID-19 during the study.
Measure: Number; unit: percentage of patients
Arm/Group | Healthcare Workers - Control | Healthcare Workers - PVP-I | Inpatients - Control | Inpatients - PVP-I | Community - Control | Community - PVP-I
Number analyzed (Participants) | 0 | 0 | 17 | 14 | 0 | 0
percentage of patients |  |  | 0 | 0 |  |

3. Primary Outcome: Percent of Community Participants Testing Positive for COVID-9.
Description: Percent of community participants that become positive for COVID-19 during the study.
Time Frame: 3 weeks
Population: Percent of community participants that become positive for COVID-19 during the study.
Measure: Number; unit: percentage of community participants
Arm/Group | Healthcare Workers - Control | Healthcare Workers - PVP-I | Inpatients - Control | Inpatients - PVP-I | Community - Control | Community - PVP-I
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 16
percentage of community participants |  |  |  |  | 0 | 0

4. Secondary Outcome: PVP-I Ease of Use
Description: Patients will rate the ease of use for PVP-I treatment on a scale from 1-5 after the initial use. Lower scores indicate increased ease of use (1="easy") while higher scores indicate increased difficulty (5="impossible").
Time Frame: 3 weeks
Population: Control groups did not receive PVP-I and therefore are excluded from the evaluation of "ease of use" of PVP-I.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthcare Workers - Control | Healthcare Workers - PVP-I | Inpatients - Control | Inpatients - PVP-I | Community - Control | Community - PVP-I
Number analyzed (Participants) | 0 | 38 | 0 | 14 | 0 | 16
units on a scale |  | 4.48 (0.80) |  | 4.43 (0.85) |  | 4.77 (0.44)

5. Secondary Outcome: PVP-I Comfort
Description: Patients will rate the comfort of PVP-I treatment on a scale from 1-5 after the initial use. Lower scores indicate increased comfort (1="not so bad") while higher scores indicate discomfort (5="worst pain of my life").
Time Frame: 3 weeks
Population: Control groups did not receive PVP-I and are therefore excluded from the analysis of "comfort" of PVP-I
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthcare Workers - Control | Healthcare Workers - PVP-I | Inpatients - Control | Inpatients - PVP-I | Community - Control | Community - PVP-I
Number analyzed (Participants) | 0 | 38 | 0 | 14 | 0 | 16
units on a scale |  | 3.25 (1.33) |  | 4.00 (1.41) |  | 3.00 (1.53)

6. Other Pre Specified Outcome: Adherence to Treatment Protocol
Description: Participants will fill out a daily questionaire assessing treatment frequency. Adherence will be calculated as the percent of correct dosing.
Time Frame: 3 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Healthcare Workers - Control | Healthcare Workers - PVP-I | Inpatients - Control | Inpatients - PVP-I | Community - Control | Community - PVP-I
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/38 | 0/17 | 0/14 | 0/2 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/38 | 0/17 | 0/14 | 0/2 | 0/16
Other Adverse Events (participants affected / at risk) | 0/11 | 0/38 | 0/17 | 0/14 | 0/2 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT04364802/Prot_ICF_001.pdf